CLINICAL TRIAL: NCT03683693
Title: Procalcitonin to Guide Antibiotic Stop in Neurocritical Care Patients. An Interventional Matched-cohort Study.
Brief Title: Procalcitonin to Guide Antibiotic Stop in Neurocritical Care Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Stoffel Lamote, Stoffel Lamote, MD, General Hospital Groeninge
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AZGS2017164
Record Dates: First submitted 2018-08-06; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Sepsis
Keywords: procalcitonin; antibiotic stewardship in ICU; Multidrug resistance; neurocritical care
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Matched cohort: historical standard of care group (patients from the period January 2016 - April 2018) versus interventional group (patients from May 2018 on)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care group (No Intervention): Historical Group = Standard of Care group. Decision for stopping antibiotics taken by ICU physician: assessment on the basis of the clinical picture and traditional inflammatory biomarkers such as crp and leucocytosis
- Procalcitonin group (Experimental): ICU physician gets on regular base PCT value, what can be used as additive tool in the decision-making for stopping antibiotics.
  Interventions: Diagnostic Test: Procalcitonin group

INTERVENTIONS:
Diagnostic Test: Procalcitonin group — The ICU physician gets on regular base (day 0, d4, d7, d11, d15, d19, d23, d27) a PCT value and the according non-binding recommendation:
  PCT < 0.5 microgram/L of 80% drop of the peak value : antibiotic stop recommended.
  PCT < 0.25 microgram/L: antibiotic stop strongly recommended. The recommendation is not-binding and can be overruled by the ICU physician. The intervention is only set up for stopping antibiotics, not for initiating. PCT measurements only happens in case of still ongoing antibiotic course. In case of a second course of antibiotics, after interruption of the initial course, new PCT measurement will take place at this point followed by the continuation of the initial schedule of PCT measurement.
  Intervention ends 28 days after inclusion.
  Arms: Procalcitonin group

SUMMARY:
Antibiotic overconsumption has been considered as one of the major contributive factors of the emergence of multidrug resistant bacteria, a serious threat particularly in intensive care units. Antibiotic stewardship programs are set up to meet this problem. Shortening the duration of antimicrobial therapy seems to be one of the strongest tools of these programs. Nevertheless, the decision to stop antibiotics in a critical care patients remains often challenging in real-life practice.

Procalcitonin (PCT), an inflammatory biomarker, has a promising profile and scores better than traditionally biomarkers as c-reactive protein (crp) and leucocytosis. Although two big multicenter randomised controlled trials showed a positive impact of PCT use in Intensive Care Unit (ICU), as it led to reduction of antibiotic exposure, the efficiency of this biomarker is still a point of debate. Notably the cost of PCT determination is a counterargument for its routinely use as it is a quite expensive test and its cost-benefit ratio has not been well studied.

The objective of this study is to test a PCT-algorithm for stopping antibiotics in a real life setting by assessing its impact on antibiotic consumption. The investigators hypothesize that it will shorten antimicrobial courses and will decrease overconsumption, with a possible positive impact on the increase of antimicrobial resistance and with no apparent adverse outcome.

DETAILED DESCRIPTION:
This is a single center, before-after, matched cohort study in a ICU of a non-university hospital. It puts the focus on neurocritical care patients as they are prone to infectious complications and these cases are often less straightforward in terms of diagnosis and management. The investigators hypothesise that such an algorithm, in addition to clinical judgement of the ICU physician, will reduce the duration of antibiotic treatment and the overall antibiotic use, could reduce selective pressure, without increase of mortality or recurrent infections.

All patients admitted to ICU with a primary non-infectious neurologic pathology will be screened for eligibility. Eligible patients can be enrolled if they meet all the inclusion criteria, there are no exclusion criteria, a matched control is available and an informed consent has provided by the patient or his or her legal representative. Patients included in the intervention group will be 1:1 matched with a patient out of the historical control group. Therefore, three fixed and two variable criteria for matching will be used. The fixed ones are: 1. pathology (traumatic brain injury; intracerebral/subarachnoid hemorrhage due to cerebral aneurysm or arteriovenous malformation; ischemic stroke; hemorrhagic stroke or other intracranial hemorrhage from; and the whether or not need for intervention (none, endovascular or neurosurgical intervention) . 2. need for mechanical ventilation within the first 12 hours after admission and 3. Glasgow coma scale (GCS) < 8 versus ≥ 8 at ICU admission or before starting sedation or anesthesia.

The two variable criteria are age (with a range of plus or minus 10 years) and the Acute Physiology and Chronic Health Evaluation (APACHE)-II score (with a range of plus or minus 15 points).

Matching will be manually, blinded for the outcome. A control group has been composed by analysing retrospectively patients admitted to our ICU from January 2016 on.

In the intervention group, doctors are additionally provided with PCT levels on regular base and with a non-binding advice on continuation or discontinuation of antibiotic therapy by electronic patient data management system feedback and by the involved microbiologist. The first PCT value will be used just as base-line, without any therapeutic consequence. Measurements will be repeated every 3-4 days, the last one is scheduled at day 27.

Patients in both groups are followed until hospital discharge, allowing assesment of hospital length of stay, hospital mortality and prevalence of multidrug resistance during hospitalisation.

Following data were collected at initiation of the trial : age, sex, BMI, pre-existing comorbidities including presence of known multidrug resistant bacteria before ICU admission, previous location before admission, reason for admission, GCS at admission to ICU, intervention, reason for antibiotic start, day of ICU admission at starting point of the study, APACHE II, the presence and type of organ dysfunction using the sequential organ-failure assessment (SOFA) score and use of mechanical ventilation.

Subsequently, following parameters will be recorded during ICU stay: SOFA score and type of organ or system failure at every PCT measurement, daily need for mechanical ventilation, source of infection when known and results of microbiological cultures. Additionally, the inflammatory biomarkers crp and leucocytosis as well as maximum temperature will be daily registered.

At the end of follow-up, every suspected infectious episode will be sorted by the investigator into four groups: 1. microbiologically documented infection (presence of a clinical and/or radiological infectious focus and pathogen identification); 2. clinically documented infection (presence of a clinical and/or radiological infectious focus, without causative pathogen identification); 3. absence of infection (absence of a clinical or radiological infectious focus) 4. possible infection (all other situations).

Data management will be performed by the investigators or research nurses. Patient's anonymity will be maintained by identifying enrolled patients of both groups with a trial identification number. The list containing the subjects name and allocation numbers are kept in strict confidence. Electronical clinical research files (CRF) or other subject related data will be protected by a password and will be put on a secured server within the hospital. Similarly, written papers (including CRF on paper) containing privacy sensitive information will be kept behind locked doors.

For the power analysis, the ICU databank has been queried, analysing the antibiotic duration of the first, uninterrupted antibiotic course of 74 patients who stayed at least 10 days in ICU in 2016 and got empirical and/or directed antibiotic therapy. A lognormal distribution with a peak value at 11.78 days has been found. After log-transformation, a mean of 2.466 with standard deviation of 0.433 was found.

The investigators aim for 20% antibiotic reduction, supported by the results of the PRORATA and the SAPS trial. This goal is ambitious, but is not unrealistic, taking into account that the study population group is traditionally characterized by high figures of antibiotic consumption. Based on these assumptions, a number of 60 patients in both groups is required for obtaining a power of 80%. This number has been increased with 10%, anticipating for patients who will die due to non-infectious reasons (pe. expected poor neurologic outcome with therapy restrictions or withdrawal) between day 7 and the end of the intervention period (day 28). In conclusion, a total of 66 patients will be included in the intervention group and will be matched with 66 patients out of the historical control group.

ELIGIBILITY:
Inclusion Criteria:

1. patients admitted to the ICU with a primary non-infectious neurological pathology:

   * Traumatic Brain Injury
   * Intracerebral Bleeding (pe. subarachnoid bleeding) due to aneurysm or arteriovenous malformation
   * Ischemic Stroke Stroke
   * Hemorrhagic stroke or other intracranial haemorrhage
   * Other non-infectious neurologic condition (as hydrocephalus, status epilepticus, postoperative complication after elective neurosurgery, ...)

   AND
2. requiring antibiotics within the first week (day 0 - day 6) after ICU-admission for a suspected bacterial infection

Exclusion Criteria:

* severe immunodeficiency and/or neutropenia: defined as (1) solid-organ transplant recipients with immunosuppressive therapy (monotherapy with corticosteroids is allowed), (2) recent chemotherapy in last 6 months, (3) hematologic malignancy with active therapy in last 2 years, (4) bone marrow transplant, (5) HIV patient with clinical complications (Pneumocystis jirovecii, Kaposi's sarcoma, lymphoma, tuberculosis, toxoplasmosis, …) or CD4 count < 200/mm3, while neutropenia has been defined as white cell count < 1000/ml.
* microbiologically proven infection with Pseudomonas, Acinetobacter baumannii, Lysteria or atypical pathogen as Chlamydia, Legionella or Mycoplasma; or Staphylococcal aureus bacteremia
* microbiologically proven meningitis or ventriculitis
* compartmentalised infection: pe. abscess, empyema
* microbiologically proven (co-)infection making a prolonged antibiotic course necessary, such as endocarditis, prosthetic joint infection or septic arthritis, osteomyelitis, chronic prostatitis, ...
* already > 24h on antibiotics before ICU admission
* (expected) ICU length of stay < 7 days
* no match available in the historical 'Standard of Care' group
* no Informed Consent obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Antibiotic use | at day 28
  We will measure the duration of the first uninterrupted antibiotic course, expressed as Days of Therapy (DOT) and as Defined Defined Daily Doses (DDD) and the Antibiotic consumption during first 28 days expressed as antibiotic free days (alive) within the first 28 days after inclusion.

SECONDARY OUTCOMES:
ICU and mortality | up to 6 months after inclusion
  We will measure ICU mortality from all causes and infection related ICU mortality by recording date of death
28-days mortality (from all causes) | at day 28
  We will measure 28-days mortality from all causes and infection related 28-days mortality by recording date of death
Hospital mortality | up to 6 months after inclusion
  date of death
ICU and hospital length of stay | up to 6 months after inclusion
  numbers of days in ICU and in hospital respectively
Duration of Mechanical ventilation | at day 28
  numbers of days alive without ventilatory support (defined as unassisted breathing) during intervention period
Recurrent infection | at day 28
  Number of patients with relapse or superinfection during ICU stay (patients requiring a new course of antibiotic therapy after a former fully completed course)
Reinfection | at day 28
  Number of patients with microbiologically proven reinfection with the same pathogen in ICU
Multidrug Resistance | up to 3 months after inclusion
  Incidence of new multidrug resistant bacteria, isolated from specimens taken for routine microbiological assessment during ICU stay
Multidrug Resistance | up to 6 months after inclusion
  Incidence of new multidrug resistant bacteria, isolated from specimens taken for routine microbiological assessment during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Stoffel Lamote, MD, Principal Investigator — AZ Groeninge
Locations (1):
- AZ Groeninge, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bell BG, Schellevis F, Stobberingh E, Goossens H, Pringle M. A systematic review and meta-analysis of the effects of antibiotic consumption on antibiotic resistance. BMC Infect Dis. 2014 Jan 9;14:13. doi: 10.1186/1471-2334-14-13. PMID 24405683
- [Background] Luyt CE, Brechot N, Trouillet JL, Chastre J. Antibiotic stewardship in the intensive care unit. Crit Care. 2014 Aug 13;18(5):480. doi: 10.1186/s13054-014-0480-6. PMID 25405992
- [Background] De Waele JJ, Schouten J, Dimopoulos G. Understanding antibiotic stewardship for the critically ill. Intensive Care Med. 2016 Dec;42(12):2063-2065. doi: 10.1007/s00134-015-4030-8. Epub 2015 Aug 20. No abstract available. PMID 26289014
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] de Jong E, van Oers JA, Beishuizen A, Vos P, Vermeijden WJ, Haas LE, Loef BG, Dormans T, van Melsen GC, Kluiters YC, Kemperman H, van den Elsen MJ, Schouten JA, Streefkerk JO, Krabbe HG, Kieft H, Kluge GH, van Dam VC, van Pelt J, Bormans L, Otten MB, Reidinga AC, Endeman H, Twisk JW, van de Garde EMW, de Smet AMGA, Kesecioglu J, Girbes AR, Nijsten MW, de Lange DW. Efficacy and safety of procalcitonin guidance in reducing the duration of antibiotic treatment in critically ill patients: a randomised, controlled, open-label trial. Lancet Infect Dis. 2016 Jul;16(7):819-827. doi: 10.1016/S1473-3099(16)00053-0. Epub 2016 Mar 2. PMID 26947523
- [Background] Iankova I, Thompson-Leduc P, Kirson NY, Rice B, Hey J, Krause A, Schonfeld SA, DeBrase CR, Bozzette S, Schuetz P. Efficacy and Safety of Procalcitonin Guidance in Patients With Suspected or Confirmed Sepsis: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 May;46(5):691-698. doi: 10.1097/CCM.0000000000002928. PMID 29271844
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Schuetz P, Balk R, Briel M, Kutz A, Christ-Crain M, Stolz D, Bouadma L, Wolff M, Kristoffersen KB, Wei L, Burkhardt O, Welte T, Schroeder S, Nobre V, Tamm M, Bhatnagar N, Bucher HC, Luyt CE, Chastre J, Tubach F, Mueller B, Lacey MJ, Ohsfeldt RL, Scheibling CM, Schneider JE. Economic evaluation of procalcitonin-guided antibiotic therapy in acute respiratory infections: a US health system perspective. Clin Chem Lab Med. 2015 Mar;53(4):583-92. doi: 10.1515/cclm-2014-1015. PMID 25581762
- [Background] Kourbeti IS, Vakis AF, Papadakis JA, Karabetsos DA, Bertsias G, Filippou M, Ioannou A, Neophytou C, Anastasaki M, Samonis G. Infections in traumatic brain injury patients. Clin Microbiol Infect. 2012 Apr;18(4):359-64. doi: 10.1111/j.1469-0691.2011.03625.x. Epub 2011 Aug 18. PMID 21851488
- [Background] Lim HB, Smith M. Systemic complications after head injury: a clinical review. Anaesthesia. 2007 May;62(5):474-82. doi: 10.1111/j.1365-2044.2007.04998.x. PMID 17448059
- [Background] Brechot N, Hekimian G, Chastre J, Luyt CE. Procalcitonin to guide antibiotic therapy in the ICU. Int J Antimicrob Agents. 2015 Dec;46 Suppl 1:S19-24. doi: 10.1016/j.ijantimicag.2015.10.012. Epub 2015 Nov 1. PMID 26607343
- See also: World Health Organisation (WHO) Collaborating Centre for Drug Statistics Methodology 2015 — http://www.whocc.no/atc_ddd_index